CLINICAL TRIAL: NCT02020928
Title: Laser Therapy Prevents Mucositis Oral in Patients Undergoing to Chemotherapy for Bone Marrow Transplantation? A Randomized Clinical Trial.
Brief Title: Laser Therapy Prevents Mucositis Oral in Chemotherapy for Bone Marrow Transplantation?
Acronym: lasertherapy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Instituto Materno Infantil Prof. Fernando Figueira (Other)
Responsible Party: Principal Investigator, Flavia orange, MD, PhD, Instituto Materno Infantil Prof. Fernando Figueira
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 3547-13
Record Dates: First submitted 2013-12-19; First posted 2013-12-25 (Estimated); Last update posted 2013-12-25 (Estimated); Status verified 2013-09

CONDITIONS: Oral Mucositis; Effects of Chemotherapy; Malignant Neoplasm of Bone Marrow
Keywords: Oral Mucositis; chemotherapy; Bone Marrow Transplantation
MeSH Terms: conditions — Stomatitis; Bone Marrow Neoplasms | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low level laser therapy (Experimental): The Low level laser therapy application is performed from the first day of conditioning of the patient until the second day after bone marrow transplantation (D + 2). The patients are divided into two groups. The first will contain the patients who will receive the red laser light, whereas the second will cover patients who receive sham or placebo controlled - the device is triggered, but not deliver the laser light.
  Interventions: Device: Low level laser therapy
- sham (Sham Comparator): patients will receive sham Low level laser therapy - the device is triggered, but not deliver the laser light
  Interventions: Device: Low level laser therapy

INTERVENTIONS:
Device: Low level laser therapy — Low level laser therapy: Laser Therapy XT (DMC) having red light with a wave length of 660 nm (± 10 nm) and infrared light with a wavelength of 808 nm (± 10 nm) is used, both power of 100 mW (± 20%), applied in a timely manner.

SUMMARY:
Setting: Oral mucositis is a very common complication of cancer treatment, accounting, often at increased risk for infections and even the interruption of treatment, interfering with the prognosis of the disease. The low intensity laser therapy has been proposed as an alternative for the treatment and prevention of this side effect, with good results in terms of clinical and functional, speeding up the process of wound healing and reducing pain.

Objective: To evaluate the effectiveness of using low power laser in the prevention of oral mucositis in patients with hematological cancer, undergoing chemotherapy for bone marrow transplantation.

Methods: There will be a Clinical Trial Randomized, double-blind study to evaluate the effectiveness of using low power laser in the prevention of oral mucositis in patients with hematological cancer, undergoing chemotherapy for bone marrow transplantation. Participate in the study, patients who are in the condition mentioned above accepting participate and have aged over 18. Will be excluded from the study patients who have autoimmune disease, which present sensitivity to laser or who have already started treatment for oral mucositis prior to this study.The study variables are:-independent variable: whether or not the red laser of low power-dependent variables: oral mucositis, degree of mucositis, chemotherapy regimen, type of blood cancer. For determining the association between the independent variable and the dependent will be used chi-square tests of association (Pearson) and Fisher's exact test, if necessary. Will calculate the risk ratio (RR) as a measure of relative risk, with the confidence interval at 95% (IC95%).Also be calculated NNT (number needed to treat to obtain benefit) and NNH (number needed to harm getting). Will be adopted a significance level of 5%. The project was approved by the Ethics and Research iMIP. All patients will be appropriately informed about the objectives of the project and will only be included if they voluntarily agree to participate by signing the consent form.

Keywords: laser, prevention and control; oral mucositis, bone marrow transplant.

DETAILED DESCRIPTION:
Inclusion Criteria: patients with blood cancers undergoing chemotherapy for

BMT; patients who agree to participate; patients older than 18 years.

Exclusion Criteria: patients with autoimmune diseases; patients who have sensitivity to the laser; patients who have already started treatment for mucositis prior to the research; HIV-positive patients.

ELIGIBILITY:
Inclusion Criteria:

* patients with hematologic cancers undergoing chemotherapy for

BMT;

* patients who agree to participate;
* patients older than 18 years.

Exclusion Criteria:

* patients with autoimmune diseases;
* patients who have sensitivity to the laser;
* patients who have already started treatment for mucositis prior to research.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2015-01; Primary Completion 2015-07 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Incidence of Oral Mucositis | From the first day after the transplantation to the eighth day after transplantation
  From the first day after the transplantation to the eighth day after transplantation

SECONDARY OUTCOMES:
Degree of mucositis | From the first day after the transplantation to the eighth day after transplantation
  From the first day after the transplantation to the eighth day after transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Flavia A de Orange, PhD, Study Director — Instituto de Medicina Integral Prof Fernando Figueira -Brazil
Locations (1):
- Instituto de Medicina Integral Prof. Fernando Figueira, Recife, Pernambuco, Brazil

REFERENCES:
- [Background] Silva GB, Mendonca EF, Bariani C, Antunes HS, Silva MA. The prevention of induced oral mucositis with low-level laser therapy in bone marrow transplantation patients: a randomized clinical trial. Photomed Laser Surg. 2011 Jan;29(1):27-31. doi: 10.1089/pho.2009.2699. Epub 2010 Oct 22. PMID 20969443